CLINICAL TRIAL: NCT03208985
Title: A Multi-Center, Open-Label Trial Investigating Behavior Related to Ella® Use in a Simulated OTC Environment (LIBRella)
Brief Title: A Study of Use of Ella®, an Emergency Contraceptive, Under Simulated OTC Conditions
Acronym: LIBRella
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 151032-001
Record Dates: First submitted 2017-06-26; First posted 2017-07-06 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Emergency Contraception
Keywords: Emergency contraception
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Use Phase (Ulipristal Acetate, 30 mg) (Experimental): One tablet of 30 mg of ulipristal acetate for emergency contraception
  Interventions: Drug: Use Phase (Ulipristal Acetate, 30 mg)

INTERVENTIONS:
Drug: Use Phase (Ulipristal Acetate, 30 mg) — All subjects enrolled in the use phase of this open-label study will be given the opportunity to purchase and take 30 mg of ulipristal acetate.
  Subjects are to use the investigational product based on their understanding of the directions on the outer packaging including Drug Facts Label and inside the product packaging (in the Consumer Information Leaflet).

SUMMARY:
This study is designed to assess whether consumers select and use ella® (ulipristal acetate 30mg), an emergency contraceptive, in a manner consistent with the OTC package directions in an OTC-like setting.

DETAILED DESCRIPTION:
All potential subject coming to a site looking to purchase EC will be offered to participate in the study. Subjects who meet the initial screening inclusion criteria for the study will review package information and make a self-selection and purchase decision. Subjects who meet all remaining inclusion criteria will purchase ella®, and use based on their understanding of the package information.

Follow-up data regarding product use and adverse events will be obtained during telephone interviews at approximately Week-2 and Week-6 after the date the subject was dispensed study product.

ELIGIBILITY:
Inclusion Criteria:

* Women who are self-pay or who are willing to be self-pay for the purposes of the study and who present for emergency contraception only for their own use

Exclusion Criteria:

* Cannot read, speak and understand English
* Cannot see well enough to read information on the label

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1270 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russel Bradford, MD, MSPH, Principal Investigator — Pegus Research, Inc.
Locations (30):
- United States (30):
  - HRA Pharma Investigational Site, Rancho Cucamonga, California
  - HRA Pharma Investigational Site, Boulder, Colorado
  - HRA Pharma Investigational Site, Denver, Colorado
  - HRA Pharma Investigational Site, Fort Myers, Florida
  - HRA Pharma Investigational Site, Miami, Florida
  - HRA Pharma Investigational Site, Orlando, Florida
  - HRA Pharma Investigational Site, Pembroke Pines, Florida
  - HRA Pharma Investigational Site, St. Petersburg, Florida
  - HRA Pharma Investigational Site, Tampa, Florida
  - HRA Pharma Investigational Site, Belleville, Illinois
  - HRA Pharma Investigational Site, Andover, Minnesota
  - HRA Pharma Investigational Site, Saint Louis Park, Minnesota
  - HRA Pharma Investigational Site, City of Saint Peters, Missouri
  - HRA Pharma Investigational Site, Kansas City, Missouri
  - HRA Pharma Investigational Site, Manchester, Missouri
  - HRA Pharma Investigational Site, St Louis, Missouri
  - HRA Pharma Investigational Site, Las Vegas, Nevada
  - HRA Pharma Investigational Site, Hackensack, New Jersey
  - HRA Pharma Investigational Site, Morristown, New Jersey
  - HRA Pharma Investigational Site, New Brunswick, New Jersey
  - HRA Pharma Investigational Site, Trenton, New Jersey
  - HRA Pharma Investigational Site, Albuquerque, New Mexico
  - HRA Pharma Investigational Site, New York, New York
  - HRA Pharma Investigational Site, Durham, North Carolina
  - HRA Pharma Investigational Site, Raleigh, North Carolina
  - HRA Pharma Investigational Site, Portland, Oregon
  - HRA Pharma Investigational Site, Bremerton, Washington
  - HRA Pharma Investigational Site, Puyallup, Washington
  - HRA Pharma Investigational Site, Seattle, Washington
  - HRA Pharma Investigational Site, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In order to be as representative as possible of the OTC EC-seeking population, when potential subjects came to a site looking to purchase EC, they've been offered the opportunity to participate in the study. If approximately 75% of subjects pass the screening criteria, self-select and both qualify and agree to purchase and enter the use phase, it was expected that up to 1270 subjects will need to be interviewed to yield 950 purchasers and 760 in use population.
Groups:
- Self-Selection Population: Subjects who accept the invitation to participate and meet study inclusion criteria, participate in a face-to-face interview at the study site and make a self-selection and purchase decision
Period: Overall Study
Arm/Group | Self-Selection Population
Started | 1270
Completed | 868
Not Completed | 402

BASELINE CHARACTERISTICS:
Population: Subjects who take at least one dose of study medication during the study.
Groups:
- Use Phase (Ulipristal Acetate, 30 mg): One tablet of 30 mg of ulipristal acetate for emergency contraception
  Use Phase (Ulipristal Acetate, 30 mg): All subjects enrolled in the use phase of this open-label study will be given the opportunity to purchase and take 30 mg of ulipristal acetate.
  Subjects are to use the investigational product based on their understanding of the directions on the outer packaging including Drug Facts Label and inside the product packaging (in the Consumer Information Leaflet).
Arm/Group | Use Phase (Ulipristal Acetate, 30 mg)
Number analyzed (Participants) | 681
Age, Continuous [Median (Full Range); unit: years] | 26.4 [14 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 681
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 173
  Not Hispanic or Latino | 506
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 224
  White | 283
  More than one race | 59
  Unknown or Not Reported | 68
Region of Enrollment [Number; unit: participants]
  United States | 681
Literacy using REALM test pr REALM Teen test [Count of Participants; unit: Participants]
  Normal Literacy | 572
  Low Literacy | 104
  Literacy Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Dosing Instances Among User Population Taken Within 120 Hours (5 Days) of Most Recent Episode of Unprotected Sex.
Description: The first primary endpoint is the proportion in which the denominator includes all dosing instances of the IP and the numerator includes all dosing instances of the IP which were taken within 120 hours (5 days) of the subject's most recent episode of unprotected sex.
Time Frame: Up to 6 Weeks
Population: User Population: subjects who have taken at least one dose of study medication during the study.
Measure: Number; unit: Dosing instances 120 hrs of unprotec.sex
Units Other Than Participants: All dosing instances
Arm/Group | Use Phase (Ulipristal Acetate, 30 mg)
Number analyzed (Participants) | 681
Number analyzed (All dosing instances) | 712
Dosing instances 120 hrs of unprotec.sex | 704

2. Primary Outcome: Proportion of Dosing Instances Among User Population in Which no More Than One Tablet Was Taken.
Description: The second primary endpoint is the proportion in which the denominator is all discrete dosing instances of the IP and the numerator includes all dosing instances where no more than one tablet was taken.
Time Frame: Up to 6 Weeks
Measure: Number; unit: Dosing no more than 1 tablet was taken
Units Other Than Participants: All dosing instances
Arm/Group | Use Phase (Ulipristal Acetate, 30 mg)
Number analyzed (Participants) | 681
Number analyzed (All dosing instances) | 712
Dosing no more than 1 tablet was taken | 712

3. Primary Outcome: Proportion of Female Selectors Who Are Not Pregnant at the Time of Selection Decision.
Description: The third primary endpoint is the proportion in which the denominator includes all females who selected to use the product (regardless of whether they purchased/used) and the numerator includes all female selectors who were not pregnant at the time of the selection decision.
Time Frame: Day 1
Population: Subjects who accepted the invitation to participate and met study inclusion criteria, participated in a face-to-face interview at the study site and made a self-selection and purchase decision, have performed an enrollment pregnancy test and either have answered 'No' to the question 'Are you currently pregnant?'
Measure: Count of Participants; unit: Participants
Arm/Group | Self-Selection Population
Number analyzed (Participants) | 819
Participants | 814

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Groups:
- Safety Population: A safety populationwas added as an analysis population, as adverse events are reportable from the time a subject signed informed consent and should thus not only be based on the user population.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/783
Serious Adverse Events (participants affected / at risk) | 15/783
Other Adverse Events (participants affected / at risk) | 132/783
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=783)
Exposure During Pregnancy (Pregnancy, puerperium and perinatal conditions) | 11 (11)
Spontaneous abortions (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Volvulus of bowel (Gastrointestinal disorders) | 1 (1)
Kidney infection (Renal and urinary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=783)
Abdominal pain lower (Gastrointestinal disorders) | 23 (23)
Nausea (Gastrointestinal disorders) | 13 (13)
Fatigue (General disorders) | 9 (9)
Urinary tract infection (Renal and urinary disorders) | 9 (9)
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Headache (General disorders) | 5 (5)
Influenza (Immune system disorders) | 5 (5)
Bacterial vaginosis (Infections and infestations) | 4 (4)
Decreased appetite (Gastrointestinal disorders) | 4 (4)
Rash (Immune system disorders) | 4 (4)
Vaginal infection (Renal and urinary disorders) | 4 (4)
Breast tenderness (Reproductive system and breast disorders) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (3)
Exposure during breast feeding (Injury, poisoning and procedural complications) | 3 (3)
Laceration (Psychiatric disorders) | 3 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (3)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dizziness (Ear and labyrinth disorders) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (2)
Sinusitis (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 2 (2)
Trichomoniasis (Psychiatric disorders) | 2 (2)
Urticaria (Immune system disorders) | 2 (2)
Vomiting (Metabolism and nutrition disorders) | 2 (2)
Vulvovaginal mycotic infection (Reproductive system and breast disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT03208985/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/85/NCT03208985/SAP_001.pdf